CLINICAL TRIAL: NCT03509688
Title: The Curative Effect and Security of Entecavir Combined Thymosin or Resveratrol on HBeAg Positive Chronic Hepatitis B Patients - a Multi-center, Random, Control, Open Clinical Trial
Brief Title: The Curative Effect of Entecavir Combined Resveratrol on HBV patients-a Multi-center, Random, Open Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Junqi Niu, MD, PhD, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3W014Q193428
Record Dates: First submitted 2017-05-02; First posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Hepatitis
Keywords: entecavir; resveratrol; thymosin; hepatitis B
MeSH Terms: conditions — Hepatitis; Hepatitis B | interventions — entecavir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- entecavir (Experimental): drug:entecavir 0.5mg/day, one time/day,144weeks
  Interventions: Drug: Entecavir
- entecavir+resveratrol (Experimental): entecavir 0.5mg/day, 144weeks intervention:resveratrol 1000mg/day, 48weeks
  Interventions: Drug: entecavir+resveratrol
- entecavir+thymosin α1 (Experimental): entecavir 0.5mg/day, 144weeks thymosin α1 2 times/week, 24weeks
  Interventions: Drug: entecavir+thymosin α1

INTERVENTIONS:
Drug: entecavir+resveratrol — entecavir+resveratrol
  Arms: entecavir+resveratrol
Drug: Entecavir — Entecavir
  Arms: entecavir
Drug: entecavir+thymosin α1 — entecavir+thymosin α1
  Arms: entecavir+thymosin α1

SUMMARY:
The purpose of this study is to use entecavir combined with other drug such as resveratrol and thymosin to treat patients with hepatitis B, which may provide a novel therapy target hepatitis B.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) infections continue to be a major public health problem worldwide. More than 400 million people worldwide are currently infected with hepatitis B virus. Approximately 20% of HBV patients will develop chronic hepatitis, and are at significant risk of developing cirrhosis or liver hepatocarcinoma. HBV is the prototype of hepadnaviridae, a family of small enveloped hepatotropic DNA viruses that can infect the liver of human.

In recent years, researches on antiviral treatment of chronic hepatitis B has made remarkable progress, interferon and nucleoside analogues which are the synthetic reverse transcriptase inhibitors can attenuate liver inflammation and fibrosis. However, HBsAg and HBeAg seroconversion ratio is merely 7% and 21%, respectively. To completely clear HBsAg is very difficult, the main reason is that HBV cccDNA (a covalently closed circular form of the viral genome through DNA repair of the relaxed circular replicative HBV DNA inside the nuclei of hepatocytes in the HBV life cycle), the template for viral and pregenomic messenger RNA cannot be eliminated, lead to the continuous replication of the virus. Apart from that, none of these therapies are completely safe and effective. Although direct antiviral therapy could efficiently control chronic active hepatitis B, drug resistance or renal toxicity could develop progressively several months after the initiation of therapy. It is thus still urgently required to identify effective anti-HBV agents.

Pegylated IFN-α (pegIFN-α) is effective in achieving sustained virologic response, defined as HBeAg seroconversion and/or hepatitis B virus (HBV) DNA levels below 20,000 copies/mL at 6 months after completion of the therapy, in only 30% of hepatitis e antigen (HBeAg)-positive and 40% of HBeAg-negative cases. However, the pegIFN-α therapy does promote HBsAg clearance or seroconversion in a small, but significant fraction of treated patients. Hence, we should develop feasible antiviral therapeutics target cccDNA in liver cells to cure chronic hepatitis B.

Resveratrol, a grape polyphenol, is representative of a group of diet-derived putative cancer chemopreventive agents encompassing, among others, curcumin, tea polyphenols and apigenin, which have attracted a lot of interest in the cancer chemoprevention community. It has shown considerable promise as a therapeutic agent in the treatment of liver ailments. Recent study found that SITR1 activators can inhibit cccDNA, and resceratrol is a member of SIRT1 activator family. Apart from that, several studies have highlighted the hepatoprotective properties of resveratrol. Resveratrol has been shown to prevent hepatic damage because of free radicals and inflammatory cytokines, induce antioxidant enzymes and elevate glutathione content. Resveratrol has also been shown to modulate varied signal transduction pathways implicated in liver diseases. For instance, resveratrol can inhibit Th17 proliferation and function, and many researches found that increasing Th17 in patients with hepatitis B. Importantly, in vitro, we found that resveratrol can significantly reduce both HBsAg and HBeAg in a dose-depend manner.

Nowadays, increasing studies focus on natural materials in the application of the treatment, and there are many health care products used resveratrol as main ingredient. Report on trial of resveratrol in healthy volunteers after daily doses of up to 5g per day administered for 29 days suggests that it is safe, as borne out by the lack of serious adverse reactions detected by clinical, biochemical or hematological analyses during the study and study follow-up. Besides, in our country, the traditional Chinese medicine also used giant knotweed (main ingredients is resveratrol) to treat viral hepatitis and autoimmune hepatitis.

Therefore, We aim to use entecavir combined with other drug such as resveratrol and peg-interferon to treat patients with hepatitis B, which may provide a novel therapy target hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* Serologic evidence of chronic hepatitis B infection more than 6 months- HBeAg positive and HBeAb negative；
* HBV DNA≥20000 IU/ml (equals to 105 copy/ml)；
* 2×ULN ≤ALT≤10×ULN，TBIL<2×ULN

Exclusion Criteria:

* Has history of decompensated liver diseases
* Has been treated with other anti-virus drugs, or anti-tumor drugs, immuno-suppression drugs
* Has a history of autoimmune hepatitis
* History of a severe seizure disorder or current anticonvulsant use
* History or other evidence of a medical condition associated with chronic liver disease other than HBV which would make the patient, in the opinion of the investigator, unsuitable for the study (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* History of thyroid disease poorly controlled on prescribed medications, elevated thyroid stimulating hormone (TSH) concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
HBeAg seroconversion rate | 48 weeks
  HBeAg seroconversion rate

SECONDARY OUTCOMES:
HBsAg loss rate, decline and seroconversion rate | 48 weeks
  HBsAg loss rate, decline and seroconversion rate
HBeAg seroconversion rate and loss rate | 72 weeks
  HBeAg seroconversion rate and loss rate
cccDNA decline level | 48 weeks
  cccDNA decline level

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, PHD, Study Chair — The First Hospital of Jilin University